CLINICAL TRIAL: NCT00356824
Title: Prospective Longitudinal Study of Interactions Between HIV and Malaria in Ugandan Children: A UCSF/Makerere University "Children With HIV and Malaria Project"
Brief Title: Relationship Between HIV and Malaria in Ugandan Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Diane V. Havlir, University of California, San Francisco
Other Study IDs: U01AI062677-01 (NIH); CHAMP
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Malaria
Keywords: Child
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Amodiaquine; Artesunate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples

GROUPS / COHORTS (1):
- 1: HIV-infected children in Uganda
  Interventions: Drug: Amodiaquine; Drug: Artesunate

INTERVENTIONS:
Drug: Amodiaquine — 200 mg oral tablet taken daily for 3 days under direct supervision at study clinic
  Other Names: Camoquin
Drug: Artesunate — 50 mg oral tablet taken daily for 3 days under direct supervision at study clinic
  Other Names: Arsumax

SUMMARY:
HIV and malaria are two of the most important diseases to afflict children in sub-Saharan Africa. However, it is unknown what relationships exist between the two diseases. The purpose of this study is to determine the relationship between HIV and malaria infections in HIV infected Ugandan children.

DETAILED DESCRIPTION:
HIV and malaria are two of the most important infectious diseases in sub-Saharan Africa. By 2000, over 25 million children and adults were living with HIV/AIDS, and 16 million people had died of the disease. Malaria is also of great importance in Africa, where over 90% of the 500 million annual cases and 2.7 million annual deaths occur primarily in children under the age of 5. Any interaction between these two diseases is of tremendous public health importance; however, data in this area, especially information on the relevance of HIV and malaria coinfection, are limited. Little is known about HIV infection's effects on antimalarial therapy, the effects of anti-HIV treatment on malaria incidence and treatment outcomes, and the effect of malaria on HIV disease progression. This study will examine HIV infected children in Uganda and evaluate these relationships between HIV and malaria.

This study will last 4 years. All participants will receive TMP/SMX as prophylaxis for malaria throughout this study. Children will be treated for all episodes of uncomplicated malaria with amodiaquine and artesunate; this treatment for malaria will be provided. Antiretroviral treatment for HIV, if deemed necessary by the study physician, will not be provided through this study. In the case of missed scheduled visits at the clinic, children and their parents or guardians will be visited at home by study staff, who will then bring the children and their parents and guardians to the clinic for their appointments.

Parents or guardians will be asked to bring children to the study clinic for all medical care. Unless instructed otherwise, the study clinic should be the only place where children in this study receive care and medications for the duration of the study. At each study visit for a new illness, children who have a temperature of 38 C (100.4 F) or greater, report having a fever in the 24 hours prior to the visit, or have suspected malaria will have their blood collected to check for malaria. If the blood is negative for malaria, the child will be treated with standard of care for the non-malaria illness in the Mulago Hospital complex.

If the blood is positive for malaria, the child will be classified as having either uncomplicated or complicated malaria. In cases of uncomplicated malaria, children will undergo medical history, a physical exam, and additional blood collection on the day of diagnosis (Day 0). Doses of amodiaquine and artesunate will be given once a day for 3 days in the study clinic by a study nurse, who will directly observe the child taking the medication. Study visits associated with uncomplicated malaria will occur on Days 1, 2, 3, 7, 14, 28, and any other day when the child feels ill; a physical exam and blood collection to check for malaria will occur at all visits. In cases of complicated malaria, children will be treated with quinine and will be referred to the Acute Care Unit of the Mulago Hospital complex.

Regardless of health during the course of the study, children will need to return to the clinic every 30 days to undergo a physical exam and blood collection to check for malaria. If malaria is found, children will undergo the 14-day standardized follow-up period as described above. At least every 3 months, additional blood collection will occur to determine HIV viral load, liver and kidney function, and immune parameters.

As of 07/01/08, all study participants with malaria will receive standard of care treatment through the Pediatric Infectious Disease Clinic. No treatment will be provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Resides within a 20 km (12.4 mi) radius of the study clinic in Kampala, Uganda
* Had a minimum of 1 regularly scheduled clinic visit in the 3 months prior to study entry
* Willing to return to the study clinic if fever or other illness occurs during this study
* Willing to avoid medications administered outside the Mulago Hospital Complex
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Intends to move more than 20 km (12.4 mi) from the study clinic during the follow-up period
* Weigh less than 5 kg (11 lbs)
* Participating in another Infectious Disease Clinic (IDC) cohort study
* Any current medical problem requiring in-patient evaluation or home care
* History of allergy or sensitivity to amodiaquine, artesunate, or quinine
* Life-threatening screening laboratory values in the absence of malaria. More information on this criterion can be found in the protocol.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-infected children in Ugana at risk for malaria infection
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V. Havlir, MD, Principal Investigator — University of California, San Francisco and San Francisco General Hospital; Moses R. Kamya, MBChB, MMed, MPH, Principal Investigator — Department of Medicine, Makerere University, Kampala, Uganda; Rukyalekere-Adeodadata Kekitiinwa, Principal Investigator — Department of Pediatrics, Makerere University, Kampala, Uganda; Anne Gasasira, Principal Investigator — Makerere University Medical School, Makerere University, Kampala, Uganda; Israel Kalyesubula, Principal Investigator — Department of Pediatrics, Makerere University, Kampala, Uganda; Grant Dorsey, Principal Investigator — University of California, San Francisco; Edwin Charlebois, Principal Investigator — University of California, San Francisco; Philip Rosenthal, Principal Investigator — University of California, San Francisco; Huyen Cao, Principal Investigator — California Department of Human Services
Locations (1):
- Pediatric Infectious Diseases Clinic, Mulago Hospital Complex, Kampala, Uganda

REFERENCES:
- [Background] Corbett EL, Steketee RW, ter Kuile FO, Latif AS, Kamali A, Hayes RJ. HIV-1/AIDS and the control of other infectious diseases in Africa. Lancet. 2002 Jun 22;359(9324):2177-87. doi: 10.1016/S0140-6736(02)09095-5. PMID 12090997
- [Background] Harms G, Feldmeier H. HIV infection and tropical parasitic diseases - deleterious interactions in both directions? Trop Med Int Health. 2002 Jun;7(6):479-88. doi: 10.1046/j.1365-3156.2002.00893.x. PMID 12031069
- [Background] Kalyesubula I, Musoke-Mudido P, Marum L, Bagenda D, Aceng E, Ndugwa C, Olness K. Effects of malaria infection in human immunodeficiency virus type 1-infected Ugandan children. Pediatr Infect Dis J. 1997 Sep;16(9):876-81. doi: 10.1097/00006454-199709000-00011. PMID 9306483
- [Background] Rowland-Jones SL, Lohman B. Interactions between malaria and HIV infection-an emerging public health problem? Microbes Infect. 2002 Oct;4(12):1265-70. doi: 10.1016/s1286-4579(02)01655-6. PMID 12467769